CLINICAL TRIAL: NCT00208936
Title: Phase II Study of Pre-Operative Chemotherapy With Taxol, Cisplatin, and 5-Fluorouracil Followed by G-CSF in Patients With Resectable Local-Regional Carcinoma of Esophagus
Brief Title: Phase II Study of Pre-Operative Chemotherapy in Patients With Resectable Local-Regional Carcinoma of Esophagus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Nabil F. Saba, Associate Professor, Emory University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0691-1995
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Esophageal Diseases
Keywords: Esophageal Diseases
MeSH Terms: conditions — Esophageal Diseases | interventions — Paclitaxel; Cisplatin; Fluorouracil; Granulocyte Colony-Stimulating Factor

INTERVENTIONS:
Drug: Taxol, Cisplatin, 5-Fluorouracil, G-CSF

SUMMARY:
This study is designed pre-operative for patients with resectable, local-regional carcinoma of the esophagus.

DETAILED DESCRIPTION:
This study is designed for patients with resectable, local-regional carcinoma of the esophagus. In a pre-operative setting, chemotherapy with Taxol, Cisplatin, and 5-Fluorouracil will be administered followed by G-CSF.

ELIGIBILITY:
Inclusion Criteria:

* Measurable disease with resectable local-regional carcinoma of the esophagus. 18 years of age or older.

Exclusion Criteria:

* Pregnant or lactating. Non-resectable local-regional carcinoma of the esophagus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 1996-01; Primary Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fanucchi, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States